CLINICAL TRIAL: NCT03957096
Title: A Phase 1 Study of SGN-CD47M in Patients With Advanced Solid Tumors
Brief Title: A Safety Study of SGN-CD47M in Patients With Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor decision based on portfolio prioritization
Sponsor: Seagen Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SGN47M-001
Record Dates: First submitted 2019-05-17; First posted 2019-05-21 (Actual); Last update posted 2020-09-17 (Actual); Status verified 2020-09

CONDITIONS: Soft Tissue Sarcoma; Colorectal Cancer; Head and Neck Squamous Cell Carcinoma; Non-small Cell Lung Carcinoma; Breast Carcinoma; Ovarian Carcinoma; Exocrine Pancreatic Carcinoma; Gastric Carcinoma; Melanoma
Keywords: HNSCC; NSCLC
MeSH Terms: conditions — Sarcoma; Colorectal Neoplasms; Squamous Cell Carcinoma of Head and Neck; Carcinoma, Non-Small-Cell Lung; Breast Neoplasms; Ovarian Neoplasms; Stomach Neoplasms; Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- SGN-CD47M (Experimental)
  Interventions: Drug: SGN-CD47M

INTERVENTIONS:
Drug: SGN-CD47M — SGN-CD47M administered intravenously

SUMMARY:
This trial will study SGN-CD47M to find out whether it is an effective treatment for different types of solid tumors and what side effects (unwanted effects) may occur. The study will have two parts. Part A of the study will find out how much SGN-CD47M should be given for treatment and how often. Part B of the study will use the dose found in Part A and look at how safe and effective the treatment is.

DETAILED DESCRIPTION:
This is a dose-escalation study designed to evaluate the safety, tolerability, pharmacokinetics (PK), and antitumor activity of SGN-CD47M in adults with advanced solid tumors. The study will be conducted in 2 parts:

Part A - Dose escalation: Up to approximately 25 patients will be treated to evaluate the safety, tolerability, and PK of SGN-CD47M, and to identify the maximum tolerated dose (MTD) and/or optimal dose.

Part B - Dose expansion: Up to approximately 180 patients will be treated in expansion cohorts at the MTD or optimal dose to further characterize the safety, PK, and antitumor activity of SGN-CD47M.

In eligible patients, standard therapies must have failed, been intolerable, or been considered medically inappropriate by the investigator. If the MTD is not reached in Part A, safety, PK, pharmacodynamic, and biomarker analyses, as well as preliminary antitumor activity, will be used to determine the optimal dose. Patients in Part A may continue on treatment until confirmed progressive disease (PD) or unacceptable toxicity, whichever occurs first. The dose(s) to be examined in Part B will be at or below the MTD and/or the optimal dose determined in Part A.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed metastatic or unresectable solid malignancy within one of the following indications:

  1. Soft tissue sarcoma
  2. Colorectal carcinoma
  3. Non-small cell lung carcinoma
  4. Head and neck squamous cell carcinoma
  5. Breast carcinoma
  6. Ovarian carcinoma
  7. Exocrine pancreatic adenocarcinoma
  8. Gastric carcinoma
  9. Melanoma
* Relapsed, refractory, or progressive disease with no appropriate standard therapy available at the time of enrollment
* ECOG performance status of 0 or 1
* Measureable disease per the Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 at baseline
* Patients of childbearing potential may not be pregnant, must agree not to become pregnant until at 30 days after last dose of study drug, and must use 2 effective means of birth control.
* Patients who can father children must use 2 effective means of birth control and must agree not to donate sperm until at least 60 days after last dose of study drug.

Exclusion Criteria:

* History of another malignancy within 3 years prior to first dose of study drug (exceptions for malignancies with negligible risk of metastasis)
* Previous exposure to CD47 or SIRPα targeted therapy
* Chemotherapy, systemic radiotherapy, biologics, other anti-neoplastic or investigational agents, and/or other antitumor treatment with immunotherapy that is not completed 4 weeks prior to first dose of SGN-CD47M. Focal radiotherapy that is not completed 2 weeks prior to the first dose of SGN-CD47M
* Known active central nervous system metastases
* Positive for hepatitis B, active hepatitis C infections, positive for human immunodeficiency virus (HIV), or known active or latent tuberculosis
* History of sickle cell anemia, auto-immune hemolytic anemia, or idiopathic thrombocytopenic purpura
* Carcinomatous meningitis
* Red blood cell transfusion within 4 weeks prior to enrollment or platelet transfusion within 2 weeks prior to enrollment
* Any active Grade 3 or higher viral, bacterial, or fungal infection within 2 weeks prior to first dose
* History of a cerebral vascular event, unstable angina, myocardial infarction, or cardiac symptoms consistent with New York Heart Association Class III-IV within 6 months prior to first dose
* Condition requiring systemic treatment with corticosteroids or other immunosuppressive medications within 2 week prior to first dose
* Active autoimmune disease, autoimmune-related toxicity from prior immuno-oncology-based therapy
* Estimated life expectancy of less than 12 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2019-07-17 (Actual); Primary Completion 2020-09-14 (Actual); Study Completion 2020-09-14 (Actual)

PRIMARY OUTCOMES:
Number of patients with adverse events | Up to approximately 24 months
Number of patients with laboratory abnormalities | Up to approximately 24 months
Number of patients with dose-limiting toxicities (DLTs) | 28 days

SECONDARY OUTCOMES:
Objective response rate (ORR) per RECIST v1.1 | Up to approximately 2.5 years
  Defined as the proportion of patients with CR or PR
ORR per iRECIST | Up to approximately 2.5 years
  Defined as the proportion of patients with iCR or iPR
Duration of objective response (DOR) per RECIST v1.1 | Up to approximately 2.5 years
  Defined as the time from start of the first documentation of objective tumor response (CR or PR) to the first documentation of disease progression or to death due to any cause, whichever comes first
DOR per iRECIST | Up to approximately 2.5 years
Duration of complete response (CR) per RECIST v1.1 | Up to approximately 2.5 years
  Defined as the time from start of the first documentation of objective tumor response to the first documentation of confirmed tumor progression or to death due to any cause, whichever comes first for the subgroup of patients achieving a CR
Duration of CR per iRECIST | Up to approximately 2.5 years
Progression-free survival (PFS) per RECIST v1.1 | Up to approximately 2.5 years
  Defined as the time from start of study treatment to first documentation of disease progression or to death due to any cause, whichever comes first
PFS per iRECIST | Up to approximately 2.5 years
Overall survival (OS) | Up to approximately 4 years
  Defined as the time from the start of any study treatment to the date of death due to any cause
Area under the concentration-time curve (AUC) | Up to approximately 24 months
Maximum concentration (Cmax) | Up to approximately 24 months
Time to Cmax (Tmax) | Up to approximately 24 months
Trough concentration (Ctrough) | Up to approximately 24 months
Incidence of antidrug antibodies (ADA) | Up to approximately 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael Schmitt, MD, PhD, Study Director — Seagen Inc.
Locations (5):
- United States (5):
  - Case Western Reserve University / University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Providence Portland Medical Center, Portland, Oregon
  - Tennessee Oncology-Nashvilee/Sarah Cannon Research Institute, Nashville, Tennessee
  - MD Anderson Cancer Center / University of Texas, Houston, Texas
  - NEXT Oncology, San Antonio, Texas